CLINICAL TRIAL: NCT05050370
Title: A Brief SMART Exercise With Chat-based Instant Messaging Personalised Support Intervention
Brief Title: A Brief SMART Exercise Instant Messaging Support Intervention - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Assistant professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UW20-019
Record Dates: First submitted 2021-01-23; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Cancer; Lung
Keywords: Lifestyle modification; physical activity; e-messages
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The experimental group will receive a face-to-face group session and a package of information on lifestyle-integrated exercise and physical activity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle-integrated exercise and care support (Experimental): The experimental group will receive a face-to-face group session and a package of instant messages related to lifestyle-integrated exercise and cancer-related information with personalized support.
  Interventions: Behavioral: Brief messaging and personalized support

INTERVENTIONS:
Behavioral: Brief messaging and personalized support — Patients will receive (i) a face-to-face group session and a package of instant messages related to lifestyle-integrated exercise (including breathing, balance, aerobic, strength, stretching exercises), cancer-related care information and support.

SUMMARY:
Lung cancer is one of the most common cancer diseases, globally and locally. Several health benefits of increased physical activity (PA) have been reported for people with cancer. PA plays a critical role across the cancer trajectory, from prevention through to post-diagnosis and has been proposed as an alternative for improving physical and psychosocial health outcomes, reducing cancer recurrence, and cancer-specific and all-cause mortality. Although there are a variety of exercise intervention programs for cancer patients, those programs were quite intensive, requiring individuals to commit extra time and effort. Feeling of overwhelmed appointments, lack of time, other barriers, including high cost and limited access to facilities are the most frequently reported barriers that prevent people from starting and maintaining exercise. Hence, the investigators propose to use a brief messaging lifestyle modification intervention program to incorporating simple and easy-to-do patient-centred home-based lifestyle-integrated exercise into daily activities of patients with lung cancer. The aims are to explore the feasibility of using instant messaging to enhance physical activity and improve their fatigue, emotion and quality of life, and obtain feedback from patients for intervention and study design improvement.

DETAILED DESCRIPTION:
Lung cancer is one of the most common cancer, globally and locally. Patients with lung cancer are in a uniquely challenging situation in their disease, comorbidities, and treatment that may lead to worsened symptoms and many negative health consequences, including fatigue, irritability, and impaired daytime functioning. Physical activity (PA) is defined as 'any bodily movement produced by skeletal muscle that results in energy expenditure'. Several health benefits of increased PA have been reported for people with cancer. PA plays a critical role across the cancer trajectory, from prevention through to postdiagnosis and has been proposed as an alternative for improving physical and psychosocial health outcomes, reducing cancer recurrence, and cancer-specific and all-cause mortality. Although there are a variety of exercise intervention programs for cancer patients, those programs were quite intensive, requiring individuals to commit extra time and effort. Most clinicians underutilise exercise therapy, regardless of its low-cost way to improve symptoms and potential health outcomes. Feeling of overwhelmed appointments, lack of time, other barriers, including high cost and limited access to facilities are the most frequently reported barriers that prevent people from starting and maintaining exercise. Low motivation, fear to exercise, lack of knowledge about benefits are the most common barriers of engaging in physical activity for cancer patients.

Hence, the current proposal is to use a brief messaging lifestyle modification intervention program to incorporating simple and easy-to-do patient-centred home-based lifestyle-integrated exercise (light to moderate physical activity) into daily activities of patients with lung cancer.

The aims are to explore the feasibility of using instant messaging to enhance physical activity and improve their fatigue, emotion and quality of life, and obtain feedback from patients for intervention and study design improvement.

ELIGIBILITY:
Inclusion criteria

* Aged 18 years and above;
* Diagnosis of non-small cell lung cancer or small cell lung cancer
* Fatigue symptom score ≥4 out of 10
* Self-reported engagement of <150 minutes of moderate-intensity PA each week
* Ambulatory and capable of all self-care activities
* Either undergoing or finished oncology therapy and/or support care
* Mentally, cognitively and physically fit to join the trial
* Able to speak and read Chinese;
* Willing to complete the patient-reported outcome questionnaire
* Completion of the Physical Activity Readiness Questionnaire
* Possession of a smartphone with instant messaging functions such as WhatsApp or WeChat.

Exclusion criteria

* Those preparing for lung operation
* Skeletal fragility
* Serious active infection
* Inability to walk
* Severe respiratory insufficiency
* Uncontrolled pain
* Diagnosed psychiatric illness such as major depressive disorder

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue level at 6 week | Baseline and 6 weeks
  measured by Functional Assessment of Cancer Therapy - Fatigue subscale, the higher scores, the more fatigue.

SECONDARY OUTCOMES:
Change in Anxiety and depressive symptoms at 6 weeks | Baseline and 6 weeks
  measured by Hospital Anxiety and Depression Scale, Each item is answered on a 4-point scale (0-3). The scores for the seven questions on depression are added together to obtain a score ranged from 0 to 21. The higher score the more depressed. The scores for the seven questions on anxiety are added together to obtain a score ranged from 0 to 21. The higher score the more anxiety and depression symptoms.
Change in sleep quality at 6 weeks | Baseline and 6 weeks
  measured by the Pittsburgh sleep quality index . The higher the score, the worse the quality.
Change in Health-related quality of life at 6 weeks | Baseline and 6 weeks
  measured by the European Organization for Research and Treatment of Cancer and Lung Module. The higher scores the worse the quality.
Change in Subjective Happiness at 6 weeks | Baseline and 6 weeks
  measured by Subjective Happiness Scale. The higher scores the more happy.
Change in Pain at 6 weeks | Baseline and 6 weeks
  measured by a question with a scale from 0 to 10; a score of "0" indicates no pain at all, a score of "10" indicates severe pain. The higher score, the more pain.
Change in dyspnea at 6 weeks | Baseline and 6 weeks
  measured by a question with a scale from 0 to 10; a score of "0" indicates no dyspnea at all, a score of "10" indicates severe dyspnea. The higher score, the more dyspnea.
Change in activity level at 6 weeks | Baseline and 6 weeks
  measured by pedometer
Change in hand grip strength at 6 weeks | Baseline and 6 weeks
  measured by a dynamometer
Change in balance at 6 weeks | Baseline and 6 weeks
  measured by single leg stand test
Change in flexibility at 6 weeks | Baseline and 6 weeks
  measured by chair sit and reach test
Change in sleep quality with objective measurement at 6 weeks | Baseline and 6 weeks
  measured by activity monitor on duration of sleep and awake intervals
Change in physical activity level with objective measurement at 6 weeks | Baseline and 6 weeks
  measured by accelerometer on the daily walking steps

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Lai, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
For those who want the patients data, please contact PI directly by written email.

REFERENCES:
- [Background] Gopalakrishnan S, Takemoto L. Binding of actin to lens alpha crystallins. Curr Eye Res. 1992 Sep;11(9):929-33. doi: 10.3109/02713689209033490. PMID 1424733
- [Background] Peddle-McIntyre CJ, Singh F, Thomas R, Newton RU, Galvao DA, Cavalheri V. Exercise training for advanced lung cancer. Cochrane Database Syst Rev. 2019 Feb 11;2(2):CD012685. doi: 10.1002/14651858.CD012685.pub2. PMID 30741408
- See also: American Lung Association - Lung Cancer — https://www.lung.org/lung-health-diseases/lung-disease-lookup/lung-cancer/resource-library